CLINICAL TRIAL: NCT01549405
Title: Ultrasound-Guided Intercostal Nerve Block for Postoperative Pain Relief in Percutaneous Nephrolitotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, derya özkan, Consultant of Anesthesiology ,MD, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: Diskapi
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-04

CONDITIONS: Nerve Block, Intercostal Nerve
Keywords: percutanous nephrolitotomy,intercostal nerve block, Ultrasound

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Control group: Group that without intercostal nerve block
- nerve block (Experimental): Group that performing intercostal block
  Interventions: Other: İntercostal nerve block

INTERVENTIONS:
Other: İntercostal nerve block — Nerve block group was administered two levels intercostal block (11 and 12th ribs) with 0.5% bupivacaine with epinephrine before surgery.
  Arms: nerve block

SUMMARY:
Percutaneous nephrolitotomy (PCNL)is an endourological procedure for the management of patients with renal calculi. Postoperative pain around the surgical area and the nephrostomy tube can being a problem. We hypothesized that intercostal nerve block at 11th and 12th rib level would alleviate postoperative pain and reduce analgesic consumption.

DETAILED DESCRIPTION:
Patients admitted for the removal of renal stones by PCNL will included in this study.Primary outcome measure will be analgesic (tramadol )consumption and visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for the removal of renal stones by percutaneous
* nephrolithotomy (PCNL)
* ASA I-II status

Exclusion Criteria:

* Respiratory or cardiac disfunction
* Neuropathy
* Coagulopathy
* BMI (Body mass index)over 30

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derya Özkan, MD, Study Director — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 1. Anesthesiology Clinic; Taylan Akkaya, MD, Principal Investigator — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 1. Anesthesiology Clinic; Emine Arık, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 1. Anesthesiology Clinic; Zeynep Koç, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 1. Anesthesiology Clinic; Nihat Karakoyunlu, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 3. Urology Clinic; Haluk Gümüs, MD, Study Chair — 1Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 1. Anesthesiology Clinic; Hamit Ersoy, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 3. Urology Clinic; Julide Ergil, MD, Study Chair — Ministry of health Diskapi Yıldirim Beyazit Training and Research Hospital 1. Anesthesiology Clinic
Locations (1):
- Derya Özkan, Ankara, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Groups:
- Nerve Block: Group that performing intercostal block
  İntercostal nerve block : Nerve block group was administered two levels intercostal block (11 and 12th ribs) with 0.5% bupivacaine with epinephrine before surgery.
Period: Overall Study
Arm/Group | Control Group | Nerve Block
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Nerve Block | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 57.3 (7.4) | 53 (13.6) | 55.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 14 | 13 | 27
Region of Enrollment [Number; unit: participants]
  Turkey | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Analgesic (Tramadol) Consumption
Description: Total consumption of tramadol will be measured for the first 24 hours.
Time Frame: Postoperative 24th hour
Reporting Status: Not Posted

2. Secondary Outcome: Postoperative Pain Will be Evaluated.
Description: The pain score (VAS)(visual analog scale) will be evaluated for the first 24 hours.("0" no pain, to "10", the maximum pain )Pain score less then 4 is acceptable.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Control: Group that without intercostal nerve block
Arm/Group | Control | İntercostal Nerve Block
Number analyzed (Participants) | 20 | 20
units on a scale | 3 [2 to 4] | 1 [0 to 3]
Statistical Analysis 1: Comparison: Control vs İntercostal Nerve Block; Test type: Superiority or Other; p = 0.002, Mann-Whitney U test

3. Primary Outcome: Total Consumption of Tramadol Will be Measured for the First 24 Hours
Time Frame: Postoperative 24th hour
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Control Group | Nerve Block
Number analyzed (Participants) | 20 | 20
mg | 199.7 (97.5) | 77.6 (39.5)
Statistical Analysis 1: Comparison: Control Group vs Nerve Block; Test type: Superiority or Other; p = 0.000, t-test, 2 sided; Mean Difference (Net) = 122.1, 95% CI 2-sided [52.98 to 132.4], Standard Deviation 58

ADVERSE EVENTS:
Arm/Group | Control | İntercostal Nerve Block
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=20) | İntercostal Nerve Block (N=20)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No